CLINICAL TRIAL: NCT07100470
Title: Metabolic Characterization of Alzheimer's Disease and Frontotemporal Dementia by 23Na-MRI and FDG-PET
Acronym: MetaAD_FTD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D25 A012
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: FTD; AD; Healthy Controls

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Diagnostic Test: Sodium MRI

INTERVENTIONS:
Diagnostic Test: Sodium MRI — Sodium MRI is used to detect early metabolic alterations in neurodegenerative diseases

SUMMARY:
Alzheimer's disease (AD) and frontotemporal dementia (FTD) are the most common forms of neurodegenerative dementia. However, their differential and timely diagnosis can be challenging for clinicians, therefore often closing the door for an early and possibly successful treatment before irreversible cerebral damage occurs. Hence, treatment options often become available only at a late point in time. In Alzheimer's disease, early neuroimaging markers are glucose hypometabolism and Amyloid-/Tau-depositions (PET). Recent findings from sodium magnetic resonance imaging (23Na-MRI) point to brain tissue sodium concentration as a metabolic marker of AD progression. Sodium is crucial for neurotransmission and cellular homeostasis maintained by the cellular Na+/K+-ATPase, depending on Adenosine-Triphosphate as energy source from the mitochondrial respiratory chain, also interacting with tau and amyloid. In this project, we aim to characterize disease-specific metabolic patterns in AD vs. FTD by performing 23Na-MRI in association to FDG-PET to support early positive and differential diagnosis and therapeutic follow-up in both diseases in association to clinical parameters such as CSF/blood markers and neuropsychological assessment. Assessment of 7T MRI including 23Na-MRI, 31P-MRS and 1H-MRI is planned with analysis of results in association with FDG-PET, Amyloid- and Tau-PET, blood and CSF biomarkers as well as neuropsychological and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Alzheimer's disease

  * CDR (Clinical Dementia Rating Scale) = 0.5 or 1
  * Progressive amnestic syndrome, associated or not with other cognitive impairments
  * Biological criteria: CSF biomarkers suggestive of AD-continuum (Jack et al., 2018)
* Patients with FTD

  * Modifications of the personality and the social conducts in the foreground (behavioral variant) (Rascovsky et al., 2011)
  * Primary progressive aphasia (Gorno-Tempini et al., 2011):

    * Effortful, agrammatic speech plus at least one of: a) impaired grammar/sentence comprehension with relatively preserved single word comprehension, or b) groping, distorted speech production (apraxia of speech)
    * Semantic language disorders
  * Compatible brain imaging: profile of atrophy and/or hypometabolism on FDG-PET (or hypoperfusion on SPECT) compatible with the diagnosis of FTD and/or absence of atypia
  * Biological criteria: No AD profile on CSF biomarkers if available; if CSF not available: diagnosis based on clinical criteria left to the judgment of the investigators
* Cognitively healthy controls

  * Absence of known psychiatric disorder
  * Score on the Folstein Mini-Mental State Examination (MMSE > or = 27) with no more than one word missing
  * Normal neuropsychological assessment for the age and the educational level, particularly Scores on the Free and Cued Selective Reminding Test (FCSRT) of >25 for free recall and >44 for total recall.

Exclusion Criteria:

* Subject with an evolving and/or badly checked psychiatric pathology (left to the judgment of the investigator).
* Subject with a grave, severe or unstable pathology (left to the judgment of the investigator) the nature of which can interfere with the variables of evaluation.
* Epileptic subjects, with poor tolerance to MRI (1.5T, 3T or 7T),
* Subject presenting contraindications to the MRI such as Pacemaker or stimulating neurosensory or implantable defibrillator, cochlear implants, eye or cerebral ferromagnetic foreign bodies close to nervous structures, metallic prostheses, neurosurgical ventriculoperitoneal shunt valves
* Known or supposed histories (< or = 5 years) of severe alcoholism or misuse of drugs
* Vascular, inflammatory or expansive, lesion visible on the MRI which can interfere with the criteria of diagnosis.
* No health insurance
* Agitation of the patient: not cooperative or agitated patients, claustrophobic subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Tissue sodium concentration | Within 4 months after inclusion
  Metabolic and structural analysis of brain characteristics by 23Na- MRI (tissue sodium concentration - TSC) at 7T MRI
Glucose metabolism | Within 4 months after inclusion
  FDG-PET (SUVR)

IPD SHARING:
Plan to Share IPD: Undecided